CLINICAL TRIAL: NCT06696287
Title: Validity and Reliability of the the 6-minute Pegboard and Ring Test in Patients with Fibromyalgia Syndrome
Brief Title: The 6-minute Pegboard and Ring Test in Patients with Fibromyalgia Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Asst. Prof., Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-13/112
Record Dates: First submitted 2024-11-03; First posted 2024-11-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with fibromyalgia

SUMMARY:
The aim of our study is to investigate the validity and reliability of the 6-minute pegboard and ring test in patients with fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia syndrome
* Being aged 18-65
* Stable use of medication for at least 3 months or longer
* Volunteering to participate in the study

Exclusion Criteria:

* Having a musculoskeletal problem that would prevent being tested
* Having cardiopulmonary and neurological disease
* Malignancy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 years who are clinically stable and diagnosed with fibromyalgia syndrome and who are being followed up at the Rheumatology Polyclinic of the Department of Physical Medicine and Rehabilitation at Kirsehir Ahi Evran University will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Arm exercise capacity | 10 minutes
  It will be assessed by 6 minute pegboard and ring test.
Functional exercise capacity | 20 minutes
  It will be evaluated using arm ergometer test.
Hand grip strength | 5 minutes
  Will be measured using a hang grip dynamometer.

SECONDARY OUTCOMES:
Activities of daily living | 10 minutes
  It will be assessed using the Milliken Activities of Daily Living scale.Total score possible is 705. Lower scores indicate a greater degree of limitation in the ability to perform daily activities in the upper extremities.
Functional status/limitation | 5 minutes
  It will be assessed with the Revised Fibromyalgia Impact Questionnaire. The maximum number of points that can be obtained is 100. Limitation due to fibromyalgia increases with increasing scores.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Kavalci Kol, Study Chair — Kirsehir Ahi Evran University; Figen Tuncay, Study Chair — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)